CLINICAL TRIAL: NCT06718296
Title: Development of a Photographic Shoulder Scale to Assess Shoulder Movements in Daily Activities
Brief Title: Development of the Photographic Shoulder Scale
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tulay Ulku SEVIM, Master's degree graduate, Istanbul University - Cerrahpasa
Other Study IDs: uHbM3J19
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Pain
Keywords: Shoulder Pain; Photographic Assessment; Shoulder Pain Assessment Scale
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: All individuals participating in the study will sign an 'Informed Consent Form', and they will be informed about what they need to do as part of the study, what situations may arise, and any questions they have will be addressed. In the research methodology, a Patient Information Form will be used to evaluate demographic and clinical information. The ASES Scale will be used to assess shoulder pain and function, the Quick DASH will be used to measure the level of disability and functional limitations, and the SF-12 Scale will be used to assess quality of life. All scales applied to the patients will be completed within one day. The re-test of the Photographic Shoulder Scale will be conducted 7 days later. Individuals who are being followed at the Orthopedics and Traumatology Department of Başakşehir Çam and Sakura City Hospital and meet the inclusion criteria will be included in the study.

SUMMARY:
Shoulder pain is a common cause of musculoskeletal complaints that affects home and work activities, as well as quality of life. It is the third most common musculoskeletal issue after spinal and knee pathologies. The prognosis for individuals with shoulder pain can vary, with approximately 50% still reporting symptoms six months after seeking primary care. In addition to pain, functional limitations can occur, interfering with work, hobbies, and social or sports activities. A large group of patients report persistent shoulder pain with a high rate of sick leave. As a result, the total economic cost associated with shoulder pain also becomes a significant concern.

The most frequently reported clinical pathologies associated with chronic shoulder pain are rotator cuff disorders, adhesive capsulitis, and glenohumeral osteoarthritis, which collectively constitute the largest portion of all shoulder pain pathologies. Patient-reported outcome measures (PROMs) are often used to assess functional loss and disability in patients. These outcome measures provide evidence about patients' perceptions of treatment and offer data on the long-term effectiveness of interventions. For this purpose, many shoulder-specific questionnaires have been developed.

Developing a tool that uses photographs representing activities to measure how much patients struggle with daily life activities could be an important alternative for shoulder patients. An example of such a scale is the Photograph Series of Daily Activities-Short Electronic Version (PHODA-SeV), which was developed for low back pain. A different photographic scale has also been developed to assess avoidance behavior in patients with shoulder pain. Similarly, developing a specific photographic scale to assess daily life activities in patients with shoulder pain could be useful in clinical practice, as it would help patients better understand the scope of the questions.

DETAILED DESCRIPTION:
The aim of our study is to develop a photographic scale that includes daily life activities involving the shoulder to assess pain and function in patients with shoulder pain. Additionally, the study aims to evaluate the structural validity and internal consistency of the developed scale.

Hypotheses:

H0: The Photographic Shoulder Scale is not valid and reliable for individuals with shoulder pain.

H1: The Photographic Shoulder Scale is valid and reliable for individuals with shoulder pain.

In the research methodology, a Patient Information Form will be used to evaluate demographic and clinical information, along with the Photographic Shoulder Scale developed by us. Additionally, the ASES (American Shoulder and Elbow Surgeons) Scale will be used to assess shoulder pain and function, the Quick DASH scale will be used to measure the level of disability and functional limitations, and the SF-12 Scale will be used to assess quality of life.

Developing a specific photographic scale to assess daily life activities in patients with shoulder pain could be useful in clinical practice for helping patients understand the scope of thequestions. This scale could contribute to identifying the difficulties in daily activities caused by shoulder pain and assist clinicians in developing treatment plans. It may also help in identifying the disability in daily life activities due to shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with traumatic or non-traumatic shoulder pain lasting for more than 3 months

Exclusion Criteria:

* Individuals with neurological and/or rheumatological diseases
* Active local or systemic infections
* A history of cancer
* Severe visual impairments
* Patients with traumatic conditions awaiting surgery

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who are being followed at the Orthopedics and Traumatology Department of Başakşehir Çam and Sakura City Hospital and meet the inclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Photographic Shoulder Scale | 1 day
  In the rehabilitation of the upper extremity musculoskeletal system, a 4-person team consisting of physiotherapists and orthopedists with theoretical and practical experience has prepared 30 activities consisting of movements commonly used in daily life. The team asked 3 specialists, "How important do you think it is to ask patients with shoulder pain about this activity?" and removed activities that the specialists deemed inappropriate, resulting in 16 activities. Photos were taken for these activities, and a scale consisting of 16 photos was applied as a pilot test to a group of 15 patients with shoulder pain. A question was asked, "Does this photo represent the activity as described?" Feedback on the topic was gathered. A scale was also added for pain assessment, using a rating from 0 to 10.
  The designed scale consists of two sections: the first section assesses pain, and the second section contains photo-based questions measuring daily life activities.

SECONDARY OUTCOMES:
Quick DASH | 1 day
  It was designed to differentiate and assess the physical disability and symptoms in patients with musculoskeletal disorders of the upper extremity. The primary component of the questionnaire, Quick DASH, consists of 11 items, each of which is rated on a 5-point ordinal scale (17). To calculate the total DASH score, all responses are summed and averaged. This value is then subtracted by 1, multiplied by 25, and provides a total score between 0-100 (with 100 being the worst score).
SF-12 | 1 day
  The Short Form 12 (SF-12) scale will be used to assess health-related quality of life. The SF-12 is a shortened version of the SF-36 Health Quality Scale. It consists of 2 components: physical and mental health. The scale includes 12 questions that assess physical, social, and mental health. A higher score indicates a better state of health and improved quality of life, while a lower score indicates a deterioration in health.
ASES | 1 day
  The ASES (American Shoulder and Elbow Surgeons) Scale consists of two sections: pain and functionality. The pain assessment includes one question, while the functionality assessment consists of 10 questions. The pain question is rated from 0 (no pain) to 10 (the worst pain imaginable). The functionality questions use a four-point Likert scale, ranging from 0 (cannot do) to 3 (not difficult). The total score ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Crookes T, Wall C, Byrnes J, Johnson T, Gill D. Chronic shoulder pain. Aust J Gen Pract. 2023 Nov;52(11):753-758. doi: 10.31128/AJGP-04-23-6790. PMID 37935145
- [Background] Sousa CO, Nascimento JDS, Pozzi F, Kardouni JR, Michener LA. Shoulder Performance Activity Test (SPAT) for People With Shoulder Pain: Feasibility, Reliability, and Validity. Phys Ther. 2023 Mar 3;103(3):pzad006. doi: 10.1093/ptj/pzad006. PMID 37172131
- [Background] Ansanello W, Dos Reis FJJ, Tozzo MC, Zatiti SCA, Meulders A, Vlaeyen JWS, de Oliveira AS. Development of the Avoidance Daily Activities Photo Scale for Patients With Shoulder Pain. Phys Ther. 2022 Feb 1;102(2):pzab268. doi: 10.1093/ptj/pzab268. PMID 34935976